CLINICAL TRIAL: NCT05640479
Title: Pregabalin Versus Dexmedetomidine for Delirium Prevention After Cardiac Surgery: A Randomized Double-Blind Trial
Brief Title: Pregabalin Versus Dexmedetomidine for Delirium Prevention After Cardiac Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Islam Morsy, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Egypt, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 35913/10/22
Record Dates: First submitted 2022-11-26; First posted 2022-12-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-03

CONDITIONS: Pregabalin; Dexmedetomidine; Delirium
MeSH Terms: conditions — Delirium | interventions — Pregabalin; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The research solutions will be formulated by a devoted pharmacist who had no further involvement in the trial. Intraoperative and postoperative parameters will be examined by a second anesthesiologist who was unaware of group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pregabalin group (Active Comparator): patients will receive pregabalin capsules (75 mg) will be given 2 h prior to induction of anesthesia and every 12 h for 24h postoperatively by nasogastric tube or orally. Patients will receive IV saline as placebo with the same rate of dexmedetomidine.
  Interventions: Drug: Pregabalin
- dexmedetomidine group (Active Comparator): patients in the dexmedetomidine group will receive after induction of GA a bolus dose of 0.4 μg/kg dexmedetomidine (over a period of 10 to 20 min) followed by an infusion of 0.2 to 0.7 μg/kg/h. Patients will receive placebo 2 h prior to induction of anesthesia and every 12 h for 24h postoperatively by nasogastric tube or orally. If patients are hemodynamically unstable, the bolus dose will be omitted. The infusion of dexmedetomidine will be continued for a maximum period of 24 h. Dexmedetomidine infusion will be not discontinued before extubation.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Pregabalin — patients will receive pregabalin capsules (75 mg) will be given 2 h prior to induction of anesthesia and every 12 hours
  Arms: pregabalin group
Drug: Dexmedetomidine — patients will receive dexmedetomidine after induction of GA a bolus dose of 0.4 μg/kg dexmedetomidine (over a period of 10 to 20 min) followed by an infusion of 0.2 to 0.7 μg/kg/h
  Arms: dexmedetomidine group

SUMMARY:
The aim of this study is to compare the effect of perioperative administration of pregabalin versus dexmedetomidine on the prevalence and lasting duration of delirium in elderly patients after cardiac surgery.

DETAILED DESCRIPTION:
Pregabalin is a beta-isobutyl of GABA with chemical similarity to gabapentin . Pregabalin binds to the alpha-2-delta subgroup of calcium channels, thereby reducing excitatory neurotransmitter release and preventing hyperalgesia and central sensitization . Pregabalin is used as anticonvulsant but has also been used as analgesic for neuropathic pain and, lately, for postoperative pain, in an attempt to reduce opioid consumption and prevent progression to chronic pain.

Dexmedetomidine with its broad range of effects including easily controllable sedation, analgesia, and anxiolysis still enables the caring medical team to interact with the patient. It reduces the activity while still maintaining the reactivity of neurons in the locus coeruleus. Therefore, it is an appealing alternative to traditional sedatives such as propofol and benzodiazepines.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 65 years of age both genders American Society of Anesthesiologists (ASA) physical status classification II or III scheduled for cardiac surgery.

Exclusion Criteria:

* Patients who had history of psychiatric diseases; inability to communicate; previous history of POD; preoperative sick sinus syndrome.
* Allergy/sensitivity to pregabalin or dexmedetomidine.
* Severe bradycardia (heart rate <50 beat per minute).
* Second-degree or above atrioventricular block without pacemaker.
* Severe hepatic or renal insufficiency.
* Previous cardiac or thoracic surgery.
* Known diagnosis of depression or other major psychiatric diseases.
* Cognitive impairment or inability to cooperate with the study.
* Renal insufficiency, and history of substance abuse.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2024-12-03 (Actual); Study Completion 2025-01-02 (Actual)

PRIMARY OUTCOMES:
Incidence of Delirium | 24 hours postoperatively for five postoperative days
  Assessment of delirium will be performed preoperatively and postoperatively at 12-h intervals or as needed according to the patient's condition using the confusion assessment method (CAM)

SECONDARY OUTCOMES:
Sedation | 24 hours postoperatively
  Sedation level will be recorded using Sedation Agitation Scale
Length of hospital stay | One month postoperatively
  Patients will stay in hospital for one month
Pain score | 48 hours postoperatively
  Postoperative pain (using VAS) at rest and movement will be measured after extubation and at 12, 18, 24, and 48 hours after surgery The Visual Analogue Scale (VAS) measures pain intensity. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').
Postoperative opioid consumption | 48 hours postoperatively
  Patients will receive 0.05mg/kg dose of intravenous morphine given to keep pain scores less than 4
Pain score | At one month after surgery
  pain intensity at one month after surgery assessed by the Visual Analogue Scale (VAS). The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').

CONTACTS AND LOCATIONS:
Overall Officials: Doha M Bakr, MD, Principal Investigator — Lecturer of Anesthesiology; Osama M Rehab, MD, Principal Investigator — Lecturer of Anesthesiology
Locations (1):
- Tanta University, Tanta, ElGharbiaa, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be upon reasonable request from the principal investigator
Supporting Information: Study Protocol, SAP, ICF
Time Frame: for one year after completion of the study